CLINICAL TRIAL: NCT07209670
Title: Umbilical Venous Versus Peripherally Inserted Central Catheters in Neonates: A Prospective Cohort Study of Complications, Catheter Survival, and CLABSI"
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Sayed Ahmed, Principal investigator, Assiut University
Other Study IDs: venous catheters in neonates
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Peripherally Inserted Central Catheter; Umbilical Venous Catheter; CLABSI - Central Line Associated Bloodstream Infection
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UVC group: UVC Group: Neonates who received umbilical venous catheters within the first 28 days of life.
  Interventions: Procedure: umbilical venous catheters insertion
- PICC group: PICC Group: Neonates who received peripherally inserted central catheters within the first 28 days of life.
  Interventions: Procedure: peripherally inserted central catheter insertion

INTERVENTIONS:
Procedure: peripherally inserted central catheter insertion — Neonates who received peripherally inserted central catheters within the first 28 days of life.
  Groups: PICC group
Procedure: umbilical venous catheters insertion — Neonates who received umbilical venous catheters within the first 28 days of life
  Groups: UVC group

SUMMARY:
This study aims to prospectively compare umbilical venous catheters (UVCs) and peripherally inserted central catheters (PICCs) in neonates, focusing on complications, catheter survival, and central line-associated bloodstream infection (CLABSI) rates

ELIGIBILITY:
Inclusion Criteria:

* Neonates admitted to the neonatal intensive care unit (NICU) requiring central venous access.

  * Infants in whom either an umbilical venous catheter (UVC) or a peripherally inserted central catheter (PICC) was inserted for clinical indications (Parenteral nutrition, administration of intravenous medications (e.g., antibiotics, inotropes, anticonvulsants, fluids) and blood sampling for frequent labs, especially in critically ill neonates).
  * Catheter insertion performed within the first 28 days of life.

Exclusion Criteria:

* Neonates with major congenital anomalies (e.g.abdominal wall defects) that may interfere with catheter placement or outcomes.
* Insertion site infection
* Infants with severe coagulopathy or bleeding disorders contraindicating central catheter insertion.
* Neonates who received both UVC and PICC simultaneously during the same admission.
* Cases with incomplete clinical records or missing follow-up data.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates admitted to the Neonatal Intensive Care Unit (NICU) at Assiut University Children's Hospital who require central venous access for parenteral nutrition, intravenous medications, or frequent blood sampling. Participants will include infants receiving either an umbilical venous catheter (UVC) or a peripherally inserted central catheter (PICC) within the first 28 days of life
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
catheter survival time | From catheter insertion until removal (up to 28 days of life or until hospital discharge, whichever occurs first)
  Number of days each catheter remains functional and in use before removal
Central Line-Associated Bloodstream Infection (CLABSI) Incidence | During the entire catheterization period (up to 28 days of life or until hospital discharge
  Number of CLABSI events per 1,000 catheter-days, diagnosed according to CDC/NHSN criteria (positive blood culture + clinical signs of sepsis with no other source)